CLINICAL TRIAL: NCT04058951
Title: Dietary Protein Quality and Quantity: Effects of a High Protein Plant-based Diet on Proteinuria Among Patients With Nephropathy - A Randomized Cross-over Trial
Brief Title: Plant Versus Animal Dietary Protein and the Effect on Proteinuria
Acronym: NYPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Nutricia, Inc. (Industry); Nordsjaellands Hospital (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NYPRO
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Kidney Insufficiency; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Complications; Hypertension; Glomerulonephritis; Kidney Diseases; Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Complications; Hypertension; Glomerulonephritis; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Animal Protein Diet (HAPD) (Placebo Comparator): Consuming a diet high in protein primarily from animal origin.
  Interventions: Other: High Animal Protein Diet (HAPD)
- High Plant Protein Diet (HPPD) (Experimental): Consuming a diet high in protein exclusive from plant origin.
  Interventions: Other: High Plant Protein Diet (HPPD)

INTERVENTIONS:
Other: High Animal Protein Diet (HAPD) — A diet containing 2,0 g protein per kilo body weight per day from primarily animal origin. To accommodate the high protein intake, the diet is supplemented with protein powder based on beef isolate.
  Arms: High Animal Protein Diet (HAPD)
Other: High Plant Protein Diet (HPPD) — A diet containing 2,0 g protein per kilo body weight per day exclusively from plant origin. To accommodate the high protein intake, the diet is supplemented with protein powder based on soy isolate.
  Arms: High Plant Protein Diet (HPPD)

SUMMARY:
The purpose of this study is to investigate if a diet high in plant protein improves kidney function in patients with kidney insufficiency and diabetes and/or hypertension and/or glomerulonephritis. The study is a non-blinded, randomized, controlled, cross-over-design with two intervention periods of each 14 days. Between the two interventions periods there is a washout period of 14 days. The participants are randomized to start with an individualized diet plan containing either high amounts of animal protein or high amounts of plant protein.

DETAILED DESCRIPTION:
The purpose of this study is to investigate if a diet high in protein (2,0 g/kg/d) of plant origin, decreases proteinuria amongst patients with diabetes, hypertension and/or glomerulonephritis with presence of micro- or mild macro albuminuria, compared to a diet high in protein of animal origin.

Kidney insufficiency is associated with increased morbidity and mortality, decreased quality of life and large financial costs for the health care system.

Evidence suggest that the source of protein may inflect the progression of the kidney disease where soy protein has shown a positive effect on estimated glomerular filtration rate and proteinuria amongst both diabetic and non-diabetic patients with nephropathy.

The study design is a 6-week, non-blinded cluster randomized, controlled, cross-over study with two intervention periods of each 14 days. Between interventions there is a washout period of 14 days. The participants are randomized to follow either a diet high in plant protein (HPPD) or a diet high in animal protein (HAPD). The diet plans are individualized to accommodate the participants energy requirements. Given the high amount of protein in the diets they are supplemented with either soy protein powder or beef protein powder. To measure primary and secondary endpoint, the participants are instructed to collect two times 24-hour urine sample at the first baseline, after 14 days and after 42 days. Blood samples are collected at the first baseline, after 14 days, at the second baseline and after 42 days.

To gain enough statistical power a minimum of 16 participants should be included. To accommodate a drop-out rate of 25%, 20 participants should be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* UACR between 30 and 800 mg/g in minimum two spot urine samples.
* Estimated Glomerular Filtration Rate (eGFR) >30 ml/min. eGFR must have been stabil over the past 6 months defined by a maximal fluctuation in eGFR of 10 ml/min.
* Minimum 30 years of age.
* Danish speaking and writing
* No changes in blood pressure medication for the past three months.

Exclusion Criteria:

* Vegetarianism or veganism
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Urine albumin creatinine ratio (UACR) | 14 days
  The change in UACR (assessed by 2 days 24-hour urinal collection) between the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Kristensen, Dr.med, Principal Investigator — Hilleroed Hospital
Locations (1):
- Hilleroed Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No